CLINICAL TRIAL: NCT01686243
Title: Real-time Ultrasound-guided Paramedian Epidural Access: Evaluation of a Novel In-plane Transverse View Technique
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Loran Mounir Solimin, MD, M.D., The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 12-560
Record Dates: First submitted 2012-07-18; First posted 2012-09-18 (Estimated); Last update posted 2019-04-08 (Actual); Status verified 2019-04

CONDITIONS: Epidural Placement
Keywords: epidural

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- echogenic 17G tuohy needles " Pajunk TuohySono (Experimental): Epidural will be placed with the aid of ultrasound and echogenic 17G Tuohy needles (Pajunk TuohySono).
  Interventions: Other: epidural needle placement with echogenic 17G Tuohy needles (Pajunk TuohySono)
- standard epidural needles (Placebo Comparator): Epidural will be placed in standard practice with standard needles.
  Interventions: Other: standard epidural placement

INTERVENTIONS:
Other: epidural needle placement with echogenic 17G Tuohy needles (Pajunk TuohySono) — Anesthesiologist will place epidural with aid of ultrasound and placement with echogenic 17G Tuohy needles (Pajunk TuohySono)
  Arms: echogenic 17G tuohy needles " Pajunk TuohySono
Other: standard epidural placement — Anesthesiologist will place epidural within standard practice, with standard needles.
  Arms: standard epidural needles

SUMMARY:
The aim of this study is to demonstrate the feasibility of a new technique using real time ultrasound guided paramedian approach to the epidural space. This approach will use transverse view of the spine utilizing curvilinear low frequency ultrasound probe "Sonosite S nerve" and echogenic 17G tuohy needles " Pajunk TuohySono"

The investigators believe that this new technique is helpful to get the best anatomic landmark for epidural catheter placement using the real-time ultrasound.

Measurable outcomes:

* Block performance time.
* Block success rate.
* Needle Depth to epidural space

Block success rate will be measured as the rate of cases that will have successful insertion of the epidural catheter using ultrasound guidance and the case is done completely under epidural anesthesia.

All cases that will be converted to general anesthesia will be counted unsuccessful.

Other measurable outcome data that will be collected will include needle depth to the epidural space, and ultrasound measured depth to the lamina

ELIGIBILITY:
Inclusion Criteria:

* Adult Patients 30 to 80 years old at time of surgery.
* Patients in whom epidural anesthesia is planned to be used as the for surgery " Surgical epidural"

Exclusion Criteria:

* Current or recent drug abuse (within past 6 months).
* Allergy to local anesthetics
* Patient refusal.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2012-07; Primary Completion 2016-11-25 (Actual); Study Completion 2016-11-25 (Actual)

PRIMARY OUTCOMES:
Real-time ultrasound-guided paramedian epidural access: | Day 1
  Block success rate will be measured as the rate of cases that will have succesful insertion of the epidural catheter using ultrasound guidance and the case is done completely under epidural anesthesia. The aim of this study is to demonstrate the feasibility of a new technique using real time ultrasound guided paramedian approach to the epidural space. This approach will use transverse view of the spine utilizing curvilinear low frequency ultrasound probe "Sonosite S nerve" and echogenic 17G tuohy needles " Pajunk TuohySono"

CONTACTS AND LOCATIONS:
Overall Officials: Sherif Zaky, M.D., Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

REFERENCES:
- [Derived] Elsharkawy H, Saasouh W, Babazade R, Soliman LM, Horn JL, Zaky S. Real-time Ultrasound-Guided Lumbar Epidural with Transverse Interlaminar View: Evaluation of an In-Plane Technique. Pain Med. 2019 Sep 1;20(9):1750-1755. doi: 10.1093/pm/pnz026. PMID 30865772